CLINICAL TRIAL: NCT00109148
Title: A Study to Assess the Safety and Efficacy of MK0364 in Obese Patients
Brief Title: An Investigational Drug Study in Obese (Considerably Overweight) Patients (0364-006)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0364-006; 2005_011
Record Dates: First submitted 2005-04-22; First posted 2005-04-25 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Obesity
Keywords: Obesity and obesity-related medical conditions
MeSH Terms: conditions — Obesity | interventions — N-(3-(4-chlorophenyl)-2-(3-cyanophenyl)-1-methylpropyl)-2-methyl-2-((5-(trifluoromethyl)pyridin-2-yl)oxy)propanamide

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0364

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of an investigational drug in patients with obesity (considerably overweight).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are obese (considerably overweight) based on body mass index.

Exclusion Criteria:

* Patients with serious or unstable current or past medical conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2004-07; Primary Completion 2005-01 (Actual); Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Addy C, Wright H, Van Laere K, Gantz I, Erondu N, Musser BJ, Lu K, Yuan J, Sanabria-Bohorquez SM, Stoch A, Stevens C, Fong TM, De Lepeleire I, Cilissen C, Cote J, Rosko K, Gendrano IN 3rd, Nguyen AM, Gumbiner B, Rothenberg P, de Hoon J, Bormans G, Depre M, Eng WS, Ravussin E, Klein S, Blundell J, Herman GA, Burns HD, Hargreaves RJ, Wagner J, Gottesdiener K, Amatruda JM, Heymsfield SB. The acyclic CB1R inverse agonist taranabant mediates weight loss by increasing energy expenditure and decreasing caloric intake. Cell Metab. 2008 Jan;7(1):68-78. doi: 10.1016/j.cmet.2007.11.012. PMID 18177726